CLINICAL TRIAL: NCT02038179
Title: University of Alabama at Birmingham CORT Project 2: The Effects of Urate Lowing Therapy (ULT) in Inflammation, Endothelial Function, and Blood Pressure
Brief Title: Center of Research Translation (CORT) Project 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F130408004; P50AR060772 (NIH)
Record Dates: First submitted 2013-12-20; First posted 2014-01-16 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Pre-hypertension; JNC 7 Stage I Hypertension
Keywords: Pre-hypertension; JNC 7 stage I hypertension
MeSH Terms: conditions — Prehypertension | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol, Then Placebo (Experimental): Participants will be asked to take 4 weeks of allopurinol (300 mg oral per day), then will crossover (after 2-4 week washout period) and take placebo for an additional 4 weeks.
  Interventions: Drug: Allopurinol; Drug: Placebo
- Placebo, Then Allopurinol (Experimental): Participants will be asked to take 4 weeks of placebo, then will crossover (after 2-4 week washout period) and take allopurinol (300 mg oral per day) for an additional 4 weeks.
  Interventions: Drug: Allopurinol; Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Participants who received allopurinol as urate lowering therapy, at a daily dose of 300 mg once daily by mouth for a 4 week duration.
Drug: Placebo — Participants who received placebo tablet (matching Allopurinol 300 mg) daily by mouth for a 4 week duration.

SUMMARY:
We propose a novel intervention for reducing BP that could have a preferential impact in patients with hyperuricemia and gout. There is a great need for new anti-hypertensives, particularly among those with gout. The proposed study is novel in its plans to investigate the physiologic mechanisms through which urate contributes to vascular disease and by which ULT may contribute to BP reduction. Also innovative, we will: 1) determine to what extent the described benefit of lowering serum urate extends beyond the adolescent population previously studied into young adults, 2) test whether a urate-lowering approach will benefit individuals that do not yet meet the current definition of hyperuricemia and do not have gout, and 3) begin to explore potential mechanisms for the higher prevalence of hypertension among African-Americans. If successful, this work could translate to the standard of clinical care and to health care recommendations for the population as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Pre-hypertension or stage I hypertension, defined as the following after the mean of two clinic measurements:
* Systolic blood pressure (SBP) ≥ 120 and <160 or;
* Diastolic blood pressure (DBP) ≥ 80 and < 100
* Serum urate ≥ 5.0 mg/dL for men or ≥ 4.0 mg/dL for women
* Age 18-40

Exclusion Criteria:

* Any current pharmacological treatment for hypertension, including diuretics (calcium channel blockers at stable doses were later allowed)
* Estimated glomerular filtration rate < 60 mL/min/1.73m2
* Current use of any urate-lowering therapy or statins
* Prior diagnosis of gout or past use of urate-lowering therapy for gout
* Prior diagnosis of diabetes
* Pregnancy, or recent delivery or last trimester pregnancy loss more recent than 3 months
* Active smokers
* Immune-suppressed individuals including transplant recipients or current use of azathioprine.
* Leucopenia with absolute white cell count < 3000 /mL, anemia with hemoglobin < 12 g/dL, or thrombocytopenia with platelet count < 150,000/mL
* Individuals of Han Chinese or Thai descent with HLAB5801 genetic phenotype
* Serious medical condition that at investigator's judgment precludes utilization of a fixed dose of allopurinol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2014-07; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Shaffer A, Rahn E, Saag K, Mudano A, Gaffo A. Variation in serum urate levels in the absence of gout and urate lowering therapy. BMC Rheumatol. 2021 Sep 8;5(1):32. doi: 10.1186/s41927-021-00202-6. PMID 34493347
- [Derived] Gaffo AL, Calhoun DA, Rahn EJ, Oparil S, Li P, Dudenbostel T, Feig DI, Redden DT, Muntner P, Foster PJ, Biggers-Clark SR, Mudano A, Sattui SE, Saddekni MB, Bridges SL Jr, Saag KG. Effect of Serum Urate Lowering With Allopurinol on Blood Pressure in Young Adults: A Randomized, Controlled, Crossover Trial. Arthritis Rheumatol. 2021 Aug;73(8):1514-1522. doi: 10.1002/art.41749. Epub 2021 Jun 5. PMID 33779064

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a 2-4 week placebo run-in prior to assignment to study arm.
Groups:
- Allopurinol Then Placebo; Placebo Then Allopurinol: Participants will be asked to take 4 weeks of allopurinol or placebo, then will crossover to the other drug (after 2-4 week washout period) and take either allopurinol or placebo for an additional 4 weeks.
  The subjects will be randomized to receive allopurinol as urate lowering therapy (ULT), at a daily dose of 300 mg once daily by mouth or placebo. Participants will be asked to take 4 weeks of allopurinol (300 mg per day PO) or placebo, then will crossover to the other drug (after 2-4 week washout period) and take either allopurinol (300 mg per day PO) or placebo for an additional 4 weeks.
Period: Phase 1 (4 Weeks)
Arm/Group | Allopurinol Then Placebo | Placebo Then Allopurinol
Started | 52 | 47
Completed | 48 | 42
Not Completed | 4 | 5
Period: Washout (2-4 Weeks)
Arm/Group | Allopurinol Then Placebo | Placebo Then Allopurinol
Started | 48 | 42
Completed | 46 | 40
Not Completed | 2 | 2
Period: Phase 2 (4 Weeks)
Arm/Group | Allopurinol Then Placebo | Placebo Then Allopurinol
Started | 46 | 40
Completed | 44 | 38
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Overall population baseline analytics are displayed. Data were collected prior to Phase 1 of the clinical trial.
Groups:
- Overall: Participants will be asked to take 4 weeks of allopurinol or placebo, then will crossover to the other drug (after 2-4 week washout period) and take either allopurinol or placebo for an additional 4 weeks.
  Placebo: The subjects will be randomized to receive allopurinol as urate lowering therapy (ULT), at a daily dose of 300 mg once daily by mouth or placebo. Participants will be asked to take 4 weeks of allopurinol or placebo, then will crossover to the other drug (after 4 week washout period) and take either allopurinol or placebo for an additional 4 weeks.
Arm/Group | Overall
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 52
  More than one race | 2
  Unknown or Not Reported | 2
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Systolic Blood Pressure collected via in-office sphygmomanometer. Report is the mean of 2 measurements.
  mm Hg | 127 (11.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Diastolic Blood Pressure collected via in-office sphygmomanometer. Report is the mean of 2 measurements.
  mm Hg | 81.3 (9.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (7.7)
Serum urate (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 5.8 (1.2)
Flow Mediated Dilation [Mean (Standard Deviation); unit: percentage of dilation] — Population: Not all participants successfully completed flow mediated dilation testing at baseline.
  percentage of dilation
    number analyzed (Participants) | 96
    (all) | 10.3 (5.2)
high sensitivity C-reactive protein (hs-CRP) [Mean (Standard Deviation); unit: mg/L] — Population: Not all participants had successful lab draws measuring highly sensitive C-reactive protein (hs-CRP) at baseline.
  mg/L
    number analyzed (Participants) | 96
    (all) | 3.5 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Compare systolic blood pressure (SBP) captured by wearing a 24 hour ambulatory blood pressure monitor during each phase of treatment (allopurinol 300 mg/day PO or placebo). Change in systolic blood pressure is calculated by comparing SBP at the end of each treatment phase to pre-treatment values.
Time Frame: 4 weeks (pre-treatment vs. post-treatment SBP)
Population: Missing data was handled with a multiple imputations approach
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Allopurinol Phase: Participants were evaluated for primary and secondary outcomes at visits pre- and post-treatment phase. During the phase participants received 300 mg, per day (PO) of allopurinol for approximately four weeks.
- Placebo Phase: Participants were evaluated for primary and secondary outcomes at visits pre- and post-treatment phase. During the phase participants received placebo, daily (PO) for approximately four weeks.
Arm/Group | Allopurinol Phase | Placebo Phase
Number analyzed (Participants) | 99 | 99
mm Hg | -1.39 (10.0) | -1.06 (8.94)
Statistical Analysis 1: Comparison: Allopurinol Phase vs Placebo Phase; Test type: Superiority; p = 0.83, paired t-test — Intent-to-Treat Analysis using multiple imputation. Imputed Means and Imputed Standard Errors of the Mean

2. Primary Outcome: Change in Flow-mediated Arterial Vasodilation
Description: Compare endothelial function as indexed by flow-mediated arterial vasodilation (FMD) within each phase of treatment (allopurinol 300 mg/day PO or placebo). Percent (%) change in FMD is calculated by comparing FMD (%) at the end of each treatment phase to pre-treatment values.
Time Frame: 4 weeks (pre-treatment vs. post-treatment FMD Values (%))
Population: Missing data was handled with a multiple imputation approach
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Allopurinol Phase | Placebo Phase
Number analyzed (Participants) | 99 | 99
percent change | 2.5 (0.55) | -0.1 (0.42)
Statistical Analysis 1: Comparison: Allopurinol Phase vs Placebo Phase; Test type: Superiority; p < 0.001, paired t-test

3. Primary Outcome: Change in Serum Levels of High Sensitivity C-reactive Protein
Description: Serum level of high sensitivity C-reactive protein will be reported as a change during treatment phase (allopurinol 300 mg/day PO or placebo). Change in serum level of C-reactive protein is calculated by comparing serum values at the end of each treatment phase to pre-treatment levels.
Time Frame: 4 weeks (pre-treatment vs. post-treatment serum levels)
Population: Data reported is imputed for missing.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Allopurinol Phase | Placebo Phase
Number analyzed (Participants) | 99 | 99
mg/L | 0.6 (0.39) | 0.8 (0.82)
Statistical Analysis 1: Comparison: Allopurinol Phase vs Placebo Phase; Test type: Superiority; p = 0.84, paired t-test

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study from date of enrollment to study completion (e.g., 12-14 weeks).
Description: The definition of adverse event and/or serious adverse event is the same as clinicaltrials.gov.
Groups:
- Allopurinol: Participants will be asked to take 4 weeks of allopurinol or placebo, then will crossover to the other drug (after 2-4 week washout period) and take either allopurinol or placebo for an additional 4 weeks.
  The subjects will be randomized to receive allopurinol as urate lowering therapy (ULT), at a daily dose of 300 mg once daily by mouth.
- Placebo: Participants will be asked to take 4 weeks of allopurinol or placebo, then will crossover to the other drug (after 2-4 week washout period) and take either allopurinol or placebo for an additional 4 weeks.
  The subjects will be randomized to receive placebo once daily by mouth.
Arm/Group | Allopurinol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/99
Other Adverse Events (participants affected / at risk) | 12/99 | 12/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=99) | Placebo (N=99)
Increase Blood Pressure (>= 160 disastolic blood pressure or >=90 systolic blood pressure) (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hyper-defecation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Itch (General disorders) | 1 (1) | 1 (1)
Abnormal Menses (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Weight Gain (General disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) — Reduced white blood cell count
Elevated Liver Enzyme (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT02038179/Prot_SAP_ICF_000.pdf